CLINICAL TRIAL: NCT01564303
Title: Potentially Nephroprotective Effects of Carnitine and Phosphodiesterase Type 5 (PDE5) Inhibitor Agent Against Contrast Media-induced Nephropathy (CMN): A Double Blind Randomized Study
Brief Title: Nephroprotective Effects of Carnitine and (PDE5) Inhibitor Agent Against Contrast Media-induced Nephropathy (CMN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Nazareth Hospital (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor-Investigator, The Nazareth Hospital, Zaher Armaly M.D. , Head of Nephrology Department, The Nazareth Hospital, Israel
Organization: The Nazareth Hospital, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: nazh7343ctil
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Contrast Media Induced Nephropathy
Keywords: Carnitine; Phosphodiesterase type 5 (PDE5) inhibitor; Contrast Media-induced Nephropathy (CMN)
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2. Acetylcysteine group (NAC+S) , aside with the saline, will (No Intervention): 2. Acetylcysteine group (NAC+S) , aside with the saline, patients will be given orally Acetylcysteine at a dose of 600 mg twice daily, on the day before and on the day of administration of the contrast agent.
  Interventions: Drug: Acetylcysteine, Phosphodiesterase type 5 inhibitor ,Carnitine
- CAR+S , aside with the saline, carnitne will be adminstrated (Experimental): Carnitine group (Car+S), aside with the saline, patients will be administrated with 20 mg/kg carnitine over 10 minutes 2 hours prior to the administration of the contrast agent and 8 hours after CT.
  Interventions: Drug: Acetylcysteine, Phosphodiesterase type 5 inhibitor ,Carnitine
- Phosphodiesterase type 5 inhibitor group (PDE5+S), aside with (Experimental): 4. Phosphodiesterase type 5 inhibitor group (PDE5+S), aside with the saline patients will be given orally 20 mg tablets of PDE5 Tadalafil once daily 2 hours prior to the administration of the contrast agent and in the subsequent day.
  Interventions: Drug: Acetylcysteine, Phosphodiesterase type 5 inhibitor ,Carnitine
- Control group (S) will be treated without any extra agents (No Intervention): Control group ( S ) , which will be treated without any extra agents, just Saline (0.9 %) will be given I.V. at a rate of 1 ml per kilogram of body weight per hour for 12 hours before and 12 hours after administration of the contrast agent.
  Interventions: Drug: Acetylcysteine, Phosphodiesterase type 5 inhibitor ,Carnitine

INTERVENTIONS:
Drug: Acetylcysteine, Phosphodiesterase type 5 inhibitor ,Carnitine — to evaluate the effect of the above agents on Kidney functioning parameters

SUMMARY:
CIAKI is a common iatrogenic. Up to date the suggested treatments for CIAKI are partially effective and have not been approved by the Food and Drug Administration yet. The lack of effective nephroprotective drug for CIAKI, emphasizes the need not only for additional new drugs but also for new strategies that might also clarify CIAKI pathophysiology. To the best of our knowledge, the potentially beneficial effect of carnitine and PDE5 inhibitors on CIAKI prevention has not been examined, so far.

DETAILED DESCRIPTION:
Hypothesis 1: More studies are focusing now on strategies to preserve tissue mitochondria and subsequently to maintain normal organ functioning [62]. One of these strategies is the use of Carnitine. Carnitine was first described in the early beginnings of the 20th century. In humans, 75% of carnitine is obtained from diet [63], whereas the rest is synthesized from two essential amino acids, lysine and methionine in kidney, liver and brain [64]. Carnitine transports long-chain acyl groups from fatty acids into the mitochondrial matrix, so they can be broken down through β-oxidation to acytl-coenzyme-A to obtain energy balance across cell membranes of tissues that derive much of their energy from fatty acid oxidation such as cardiac and skeletal muscles [66,67].

Plasma concentration of free carnitine is in dynamic balance with acylcarnitines with the acyl to free carnitine ratio of ≤ 0.4 being considered normal [65], however, in uremic patients, this balance is disrupted, and this ratio is altered because of a larger amount of free carnitine is esterified to acyl-carnitine to "buffer" the excess of acyl groups, modulating the bound CoA to free CoA [68]. This may cause several metabolic disturbances at the cellular level, including impaired mitochondrial fatty acid oxidation and energy production, accumulation of toxic acyl moieties, and inhibition of key enzymes of metabolic pathway [69]. These metabolic abnormalities may lead to the several clinical alterations often observed in these patients, such as muscle weakness and myopathy, loss of body protein and cachexia, insulin resistance and glucose intolerance, plasma lipid abnormalities, anemia refractory to erythropoietin (EPO) treatment, cardiomyopathy, and intradialytic symptoms [70,71,72]. Thus, the imbalanced in acyl/free carnitine ratio may explain the higher risk of patients with chronic renal failure to CIAKI. However, Carnitine supplementation may contribute to the regeneration of sequestrated free CoA and to maintain normal metabolic processes [66,67].

Experimental studies shows that L-propionylcarnitine, a propionyl ester of L-carnitine, was able to prevent cyclosporine (immunosuppressive agent following organ transplantation) induced acute nephrotoxicity, reducing lipid peroxidation and significantly lowering blood pressure. L-propionylcarnitine prevented the decline in creatinine clearance in cyclosporine chronically treated animals [73]. Patients treated with carnitine displayed improved physical performance and treatment-related chronic fatigue, cardiovascular disease, cancer, diabetes, and other chronic syndromes, caused by impaired carnitine production in kidney disease [36-38]. In the last decade there are increasing reports describing the beneficial use of carnitine for a better energy metabolism (mitochondrial metabolism). Carnitine increases albumin and protein levels, restores antioxidant defenses, and improves nutritional status, cardiac, vascular smooth muscle, and muscular function [39-42]. The postulated beneficial effect of carnitine treatment is by directing lipids towards oxidation and ATP production. Another possible protective effect of carnitine on contrast media induced lesions is its ability to suppress the development of oxidative stress and free radical generation [74]. Free radicals, and in particular hydroxyl radical, lead to lipid peroxidation of cell membranes, causing degradation of phospholipids, resulting in increased production of renal vasoconstrictors [75].

It should be emphasized that carnitine is available as a medication and is approved by the FDA for treating secondary deficiency due to metabolic diseases. Intravenous administration of carnitine is safe, and its pharmacokinetics can be analyzed just by knowing the pre-dose level in plasma [76]. Further, after single-dose intravenous administration of (0.5 g) of acetyl-L-carnitine, its rapidly, but not completely hydrolyzed, and acetyl-L-carnitine and L-carnitine concentrations return to baseline within 12 hours. Even in high doses; intravenous doses as high as 300 mg/kg have been administered with no apparent toxicity. However, the most commonly reported adverse effects are few and nonserious including gastritis, diarrhea, and body odor.

The beneficial carnitine supplies have been extensively evaluated in animals and humans during the last 20 years. As a result, several experts have already aimed to revise the clinical evidence supporting its therapeutic use. In Addition to the light of the growing experimental evidences for the beneficial effects of carnitine as an antioxidant and as a beneficial modulator of mitochondrial energy expenditure, it is tempting to explore the possibility that carnitine may exert nephroprotective effects in CIAKI.

Hypothesis 2: Another new upraising strategy that has been used in attenuating renal injury in experimental studies is the use of phosphodiesterase type 5 (PDE5) inhibitor agents [77, 78]. PDE5 inhibitors are approved by the FDA for erectile dysfunction and pulmonary hypertension. The latter have been found to exert a significant antiapoptotic effect on renal tubular cells exposed to partial unilateral ureteral obstruction [79]. Part of the physiological process of PDE5 inhibition involves the release of nitric oxide (NO). Brando et al. linked the increase in available pool of cyclic 3,5 guanosine monophosphate (cGMP) by phosphodiesterases inhibitors to prevention and ameliorating chronic renal damage mainly by attenuating hypertension and retarding progression of renal disease [80]. Furthermore a PDE 5 inhibitor has been demonstrated to be able to ameliorate nephrotoxicity. Noami H. et al. have shown that FR226807, a selective PDE5 inhibitor, ameliorates cyclosporine A nephrotoxicity with further increases in cGMP content [81]. These observations may be of relevance for contrast media induced renal injury and suggest PDE5 inhibition as a potential therapeutic approach to this clinical entity.

In sum, CIAKI is a common iatrogenic. Up to date the suggested treatments for CIAKI are partially effective and have not been approved by the Food and Drug Administration yet. The lack of effective nephroprotective drug for CIAKI, emphasizes the need not only for additional new drugs but also for new strategies that might also clarify CIAKI pathophysiology. To the best of our knowledge, the potentially beneficial effect of carnitine and PDE5 inhibitors on CIAKI prevention has not been examined, so far.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of 18 years old or older
2. CKD stage 3 according to GFR-MDRD equation.
3. Two consecutive stable plasma Creatinine levels during the last 2months.
4. Elective computed tomography (CT) with a nonionic low-osmolality radiographic contrast agent.

Exclusion Criteria:

1. Acute/ chronic renal failure. Acute renal failure is defined as a change in serum creatinine concentration of at least 0.5 mg/dL, or 25% from creatinine measured before the study to that of the day of the procedure.
2. Intercurrent illness: e.g. fever… etc.
3. Recent exposure to radiographic contrast media in the last month before enrollment.
4. Allergy to contrast agents, PDE inhibitors or NAC.
5. Hypotension
6. Pregnancy and lactation
7. Multiple Myeloma
8. Intravenous diuretics therapy
9. Therapy with any of the nephroprotective drugs 2 weeks before enrollment such as N.A.C. PED5 inhibitor or Carnitine for any reason.
10. Severe Congestive Heart Failure, Acute Myocardial Infarction, moderate to severe liver failure (Child-Pugh class B or C).
11. Concomitant use of Nitrates, CYP3A inhibitors (e.g Ketonazole, Itraconazole) or Inducers (e.g Rifampin)
12. Therapy with potential nephrotoxicity such as NSAID OR COX2 Inhibitors, Aminoglycosides, and Amphotericin B, Cisplatin, etc in the last two weeks before enrollment or within 5 days following the procedure.
13. Therapy with Metformin in the last 48 hours before the procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-11 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Kidney functioning biomarker | NGAL and creatinine will be assessed before CT and 2, 6, 12,24,48,120 hours after CT
  7 time points over 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nazreth Hospital, Nazareth, Nazareth, Israel